CLINICAL TRIAL: NCT04252339
Title: Phase 1, Open Label, Dose Escalation and Expansion Study of RLY-1971, a Highly Potent and Selective SHP2 Inhibitor, in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: RLY-1971 in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO43242; REFMAL 678 (Other: Sarah Cannon Development Innovations)
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor, Unspecified, Adult
Keywords: Solid Tumors; Advanced or Metastatic Solid Tumors; Phase 1; First in Human (FIH); SHP2 inhibition; PTPN11; Bypass Resistance; GDC-1971; RO7517834
MeSH Terms: conditions — Noonan Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RLY-1971 - Dose Escalation/Expansion (Experimental): Dose Escalation: Oral dose of RLY-1971 until Maximum Tolerated Dose (MTD), and Recommended Phase 2 dose (RP2D) are identified
  Dose Expansion: Oral dose of RLY-1971 once Maximum Tolerated Dose (MTD), and Recommended Phase 2 Dose (RP2D) are identified.
  Interventions: Drug: RLY-1971

INTERVENTIONS:
Drug: RLY-1971 — RLY-1971 is an oral inhibitor of SHP2.
  Other Names: GDC-1971; RO7517834

SUMMARY:
This study is a multi-center, open-label, dose escalation and expansion study of RLY-1971 in subjects with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Dose escalation/dose expansion study to assess the MTD, safety, tolerability, PK and preliminary anti-tumor activity of RLY-1971. Approximately 70 patients

ELIGIBILITY:
Inclusion Criteria:

Subject is willing and able to provide written informed consent for the study prior to the performance of any study-specific procedures Subject is a male or female subject ≥18 years of age at the time of consent Subject must have an ECOG PS ≤ 1 Subject must have histologically or cytologically confirmed advanced or metastatic solid tumor Subjects who are refractory to FDA-approved, standard therapy or for which standard or curative therapy does not exist or is not considered sufficient or appropriate by the patient or Investigator Subject must have radiographically measurable or evaluable disease Subject must have recovered from the reversible effects of prior anti-neoplastic therapy, except for alopecia and ≤ grade 2 neuropathy.

Subject has adequate end organ function Subject is willing to comply with all protocol-required visits, assessments, and procedures Male and female subjects of child-bearing potential are willing to use medically acceptable methods of birth control from the screening visit through 30 days after the last dose of study medication

Exclusion Criteria:

Subjects with documented history of tumor mutations that may not be amenable to treatment with RLY-1971, including:

KRAS mutations: G12D, G12V, G13X, and Q61X BRAF V600E mutation MEK mutations Subjects with prior antineoplastic therapy within 3 weeks of Study Day 1, or 5 half-lives, whichever is shorter Subjects with prior palliative radiotherapy within 1 week of Study Day 1 Subjects who have had major surgery or trauma, or incomplete recovery from surgery or trauma, within 4 weeks of Study Day 1 Subjects with known central nervous system (CNS) metastases or primary CNS tumor that is associated with progressive neurologic symptoms or requires increasing doses of corticosteroids to control the CNS disease. If patient requires corticosteroids for management of CNS disease, the dose must have been stable for the 2 weeks preceding C1D1, or subject has new lesions appearing on follow up brain MRI that require CNS-directed intervention.

Subjects with a history or evidence of ophthalmic disease Subjects with a history or evidence of significant cardiac dysfunction Subjects with a history or evidence of significant gastrointestinal disease Subjects with other serious concurrent medical conditions Subject is pregnant, as documented by a serum beta human chorionic gonadotropin (β-hCG) pregnancy test consistent with pregnancy obtained within 7 days before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Escalation Phase - 18 month Enrollment
  MTD is defined as a dose level immediately below that at which ≥2 of 6 subjects experience a DLT during the first cycle.
Recommended Phase 2 Dose (RP2D) | Escalation Phase - 18 month Enrollment
  RP2D may be the same dose level or lower than the determined MTD.

SECONDARY OUTCOMES:
Plasma concentration levels of RLY-1971 | At the beginning of Cycle 1 & Cycle 2 (Each Cycle is 21 days)
  Blood samples may be taken at pre-dose, 0.5, 1, 2, 4, 6, and 8hrs on Cycle 1 Day 1 and 15, 24 hrs post dose on Cycle 1 Day 2, and pre-dose on Cycle 2 Day 1
Objective Response Rate (ORR) | Through study completion (an average of one year)
  Evaluation by RECIST 1.1; ORR is defined as the proportion of subjects in the response evaluable population who achieve the best overall response (BOR) of CR or PR
Disease Control Rate (DCR) | Through study completion (an average of one year)
  DCR is defined as the percentage of response evaluable subjects who achieve a BOR of CR, PR or SD for at least 3 months

OTHER OUTCOMES:
Changes in phospho-ERK levels | At the beginning of Cycle 1 Day 1 post and predose (Cycle = 21 days)
  Blood will be collected at pre-dose at baseline on Cycle 1, Day 1 (C1D1) and at 3 time points (pre-dose, 2 hours post-dose, and 4 hours post-dose) on Cycle 1, Day 15 (C1D15) to assess the extent of target engagement
Tumor mutations by sequencing circulating tumor DNA (ctDNA) | At the beginning of Cycle 1 Day 1
  Blood will be collected at screening and at End of Treatment on all patients
Duration of Response (DOR) | Through study completion (an average of one year)
  DOR is defined as the time from the participant's initial objective response (CR or PR) to RLY-1971, to disease progression or death due to any cause, whichever occurs first
Progression-free Survival (PFS) | Through study completion (an average of one year)
  PFS is defined as the time from the start of study treatment to the first documented disease progression per RECIST v1.1, or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (6):
  - Florida Cancer Specialist-Lake Mary, Lake Mary, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Tennessee Oncology; Sarah Cannon Research Institute, Nashville, Tennessee